CLINICAL TRIAL: NCT00000357
Title: Buprenorphine Maintenance for Opiate Dependence
Brief Title: Buprenorphine Maintenance for Opiate Dependence - 6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Pennsylvania (Other)
Purpose: Treatment
Other Study IDs: NIDA-3-0012-6; Y01-3-0012-6
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1993-12

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: opiate dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to determine the efficacy of buprenorphine as a substitution pharmacotherapy for opiate dependence.

ELIGIBILITY:
Please contact site for information.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 1992-06; Primary Completion 1993-08 (Actual); Study Completion 1993-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles O'Brien, M.D., Ph.D., Principal Investigator — PDVAMC Treatment Research Center
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States